CLINICAL TRIAL: NCT00074139
Title: A Pharmacokinetic Interaction Study Of Docetaxel (Taxotere) 75 mg/mIV On The Combination Therapy Doxorubicin (50 mg/m) And Cyclophosphamide (50 mg/m) In The Treatment Of Advanced Breast Cancer
Brief Title: Docetaxel, Doxorubicin, and Cyclophosphamide in Treating Women With Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No patients were enrolled
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CWRU040314; CDR0000343609 (Registry Identifier: PDQ (Physician Data Query)); CWRU-AVEN-1103; AVENTIS-XRP6976D/1001
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, doxorubicin, and cyclophosphamide, use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them at different times, may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective for breast cancer.

PURPOSE: Randomized phase I trial to compare the effectiveness of two regimens of docetaxel combined with doxorubicin and cyclophosphamide in treating women who have advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pharmacokinetic profile of docetaxel, doxorubicin, and cyclophosphamide in women with advanced breast cancer.

Secondary

* Compare the pharmacokinetic profile of this regimen in these patients vs the historical pharmacokinetic profile of docetaxel.

OUTLINE: This is a randomized, open-label, crossover, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive doxorubicin IV over 15 minutes and cyclophosphamide IV over 15 minutes on day 1 followed by doxorubicin IV over 15 minutes, cyclophosphamide IV over 15 minutes, and docetaxel IV over 1 hour on day 22.
* Arm II: Patients receive doxorubicin IV over 15 minutes, cyclophosphamide IV over 15 minutes, and docetaxel IV over 1 hour on day 1 followed by doxorubicin IV over 15 minutes and cyclophosphamide IV over 15 minutes on day 22.

Treatment in both arms continues in the absence of disease progression or unacceptable toxicity. Patients may receive additional therapy at the discretion of the treating physician.

Patients are followed at 3-4 weeks.

PROJECTED ACCRUAL: A total of 24 patients (12 per treatment arm) will be accrued for this study within 7 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced breast cancer

  * Adjuvant setting for high-risk disease allowed
* No symptomatic evidence or history of brain metastases
* No leptomeningeal metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 to 69

Sex

* Female

Menopausal status

* Not specified

Performance status

* WHO 0-2 OR
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count at least 2,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic

* Bilirubin less than upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN (1.5 times ULN if alkaline phosphatase greater than 2.5 times ULN)
* Alkaline phosphatase no greater than 5 times ULN

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* LVEF or shortening fraction greater than lower limit of normal by MUGA or echocardiography
* Cardiac function normal
* No congestive heart failure
* No unstable angina pectoris
* No myocardial infarction within the past year
* No uncontrolled hypertension
* No high-risk uncontrolled arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* No active uncontrolled infection
* No active peptic ulcer
* No unstable diabetes mellitus
* No other serious illness or medical condition
* No contraindication to corticosteroids
* No pre-existing grade 2 or greater motor or sensory neurotoxicity
* No psychological, social, familial, or geographical reason that would preclude study follow-up
* No history of significant neurologic or psychiatric disorder (e.g., psychotic disorder, dementia, or seizures) that would preclude understanding and giving informed consent
* No other neoplasm within the past 10 years except curatively treated nonmelanoma skin cancer, carcinoma in situ of the cervix, ipsilateral ductal carcinoma in situ of the breast, or lobular carcinoma in situ of the breast

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 6 months since prior anthracycline or taxoid (e.g., paclitaxel or docetaxel) therapy
* No prior cumulative anthracycline dose greater than 240 mg/m^2

Endocrine therapy

* Concurrent corticosteroid treatment allowed provided treatment was initiated more than 6 months before study entry and at a dose of less than 20 mg of methylprednisolone or equivalent
* No concurrent ovarian hormonal replacement therapy

Radiotherapy

* Not specified

Surgery

* More than 2 weeks since prior major surgery

Other

* More than 30 days since prior participation in another clinical trial with any investigational drug or device
* No other concurrent experimental drugs
* No other concurrent systemic anticancer therapy
* No concurrent aminoglycoside antibiotics

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-09; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth A. Overmoyer, MD, FACP, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center, Cleveland, Ohio, United States